CLINICAL TRIAL: NCT02592811
Title: Endoscopic Sphincterotomy Plus Large-Balloon Dilatation (ESLBD) Versus Conventional Endoscopic Treatment for Removal of Large Common Bile Duct Stones : A Prospective Comparative Multi Center Randomized Study
Brief Title: Comparison of Endoscopic Sphincterotomy Plus Large-balloon Dilatation and Conventional Treatment for Large CBD Stones
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, MD, Société Française d'Endoscopie Digestive
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SocieteFranceED
Record Dates: First submitted 2015-10-05; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Choledocholithiasis; Large Common Bile Duct Stone
Keywords: Cholangiopancreatography; therapeutic strategy; Endoscopic Retrograde
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde; Sphincterotomy, Endoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESLBD (Active Comparator): Endoscopic Sphincterotomy plus Large Balloon Dilatation +/- lithotripsy
  1. ERCP with deep cancellation of BDS
  2. Endoscopic large sphincterotomy
  3. Large Balloon Dilatation of Oddi Sphincter: with the HERCULES, Cook 12, 15, 18 or 20 mm of diameter (adapted to stone diameter)
  4. Stone extraction with dormia basket or extraction balloon
  5. Mechanical Lithotripsy if needed
  Interventions: Procedure: ERCP; Procedure: Endoscopic Sphincterotomy; Device: Large Balloon Dilatation of Oddi Sphincter; Procedure: Stone extraction
- CONV (Active Comparator): Conventional treatment associating Endoscopic Sphincterotomy +/- Mechanical Lithotripsy (ES+/-LM)
  1. ERCP with deep cancellation of BDS
  2. Endoscopic large sphincterotomy
  3. Stone extraction with dormia basket or extraction balloon
  4. Mechanical Lithotripsy if needed
  Interventions: Procedure: ERCP; Procedure: Endoscopic Sphincterotomy; Procedure: Stone extraction

INTERVENTIONS:
Procedure: ERCP — Common bile duct cannulation with a cannulation catheter
  Other Names: Cholangiogram with deep cannulation of CBD
Procedure: Endoscopic Sphincterotomy — Endoscopic large sphincterotomy
  Other Names: ES
Device: Large Balloon Dilatation of Oddi Sphincter — Large Balloon Dilatation : with the HERCULES, Cook 12, 15, 18 or 20 mm of diameter (adapted to stone diameter)
  Other Names: LBD, LBDS
  Arms: ESLBD
Procedure: Stone extraction — After dilatation, extraction of stones is done with dormia basket or extraction balloon and if not possible a mechanical lithotripsy is performed

SUMMARY:
Bile duct stone extraction is impossible after endoscopic sphincterotomy (ES) alone in approximatively 10% of cases (mostly because of stones' size). Adjunction of a mechanical lithotripsy (ML) is well established to improve clearance of common bile duct (CBD) stones. Because of inconstant success, high cost, and length of procedure, an alternative method was proposed in 2003: endoscopic sphincterotomy plus large balloon dilatation (ESLBD). If the safety of ESLBD is accepted in all recent published studies, it remains controversial wether ESLBD is superior to conventional endoscopic treatment associating ES± ML for CBD stones. Procedure treatment and place of ESLBD in CBD stones therapeutic strategy is unclear.

The purpose of this prospective comparative multi center randomized study is to evaluate the superiority or not of ESLBD on conventional treatment (ES±ML) for the treatment of large bile duct stone (≥13mm) after standard ES, and to propose a new CBD stones therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CBD stones with a smaller diameter ≥ 13mm on cholangiogram

Exclusion Criteria:

* Active or history of acute pancreatitis
* Presence of intrahepatic stones
* History of Billroth II or roux-en-Y reconstruction
* Coagulation disorder (partial thromboplastin time > 42 seconds, prothrombin time (Quick value) < 50% and platelet count of <50 000/mm3)
* Current anticoagulation or clopidogrel treatment
* Pregnancy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Success of common bile duct clearance in one session of ERCP (endoscopic retrograde cholangiopancreatography) | 1 month

SECONDARY OUTCOMES:
Number of patients with mild or severe BLEEDING (Morbidity) after ERCP | 1 month
  Immediate complications were noted :
  * bleeding : mild if blood transfusion not necessary, and severe if blood transfusion necessary
  * Clinical data (pain, fever, vomiting...) are noted during first month
  * Clinical examination and blood tests (Blood count, C reactive protein, lipase blood test, hepatic tests, creatininemia) were noted at the 30th day after procedure
  * In case of bleeding suspected, a new ERCP was done
  * Number of patients with bleeding and with any complication in both groups were noted and compared
Number of patients with mild or severe ACUTE PANCREATITIS (Morbidity) after ERCP | 1 month
  Immediate complications were noted :
  * Acute pancreatitis : defined by the association of abdominal pain and lipase blood test > 3 N
  * Severity of acute pancreatitis was evaluated on CT index, and on evolution data
  * Clinical data (pain, fever, vomiting...) are noted during first month
  * Clinical examination and blood tests (Blood count, C reactive protein, lipase blood test, hepatic tests, creatininemia) were noted at the 30th day after procedure
  * Abdominal CT was performed in case of suspected acute pancreatitis
  * Number of patients with Acute Pancreatitis and any complication in both groups were noted and compared
Number of patients with PERFORATION (Morbidity of ERCP) | 1 day
  * Suspected on clinical data (pain, fever, vomiting...) and blood tests (Blood count, C reactive protein) noted during first day after ERCP:
  * confirmed on CT
  * Number of patients with perforation in both groups were noted and compared, and global morbidity in both groups were noted and compared
Number of patients with post ERCP INFECTION as angiocholitis, cholecystitis or urine infection, septicemia (Morbidity of ERCP) | 1 month
  * Suspected on clinical data (pain, fever, vomiting...), blood tests (Blood count, C reactive protein, blood and urine cultures), noted during first day after ERCP, during 30th day and more if necessary in the meantime
  * Abdominal US and CT were performed if necessary
  * Number of patients with infection in both groups were noted and compared, and global morbidity in both groups were noted and compared
GLOBAL MORBIDITY of ERCP (number of patients with bleeding and/or acute pancreatistis and/or perforation and/or infection) | 1 month
  - Number of patients with any complication as bleeding, acute pancreatitis, perforation, infection (as angiocholitis, cholecystitis, urine infection or septicemia) happened in both groups during the first month after the procedure were noted and compared
MORTALITY of ERCP | 1 month
  - Number of death happened in both groups during the first month after the procedure were noted and compared
Number of patients with recurrence of BDS | 1 month
  * Clinical data (pain, fever, vomiting...) are noted during first month
  * Clinical examination and blood tests (Blood count, C reactive protein, lipase blood test, hepatic tests, creatininemia) were noted at the 30th day after procedure
  * In case of recurrence BDS suspected, abdominal US and/or CT and/or MRI and/or EUS (Endoscopic Ultrasonography) were done, and if BDS was confirmed, a new ERCP was done
  * Number of patients with recurrence of BDS in both groups in the first month after the procedure were noted and compared
Length of procedure | Day one
  For each patient, time was noted at the beginning and at the end of ERCP
Cost of procedure | Day one
  All the instrument used during ERCP (endoscopic retrograde cholangiopancreatography) for each patient were noted, and at the end of procedure cost of all instruments were recorded
comparison of the frequency of mechanical lithotripsy of both groups | Day one
  In both groups mechanical lithotripsy can be performed in case of impossibility of stone extraction. The rate of lithotripsy performed in both groups were compared

CONTACTS AND LOCATIONS:
Overall Officials: David KARSENTI, MD, Principal Investigator — Société Française d'Endoscopie Digestive

REFERENCES:
- [Derived] Karsenti D, Coron E, Vanbiervliet G, Privat J, Kull E, Bichard P, Perrot B, Quentin V, Duriez A, Cholet F, Subtil C, Duchmann JC, Lefort C, Hudziak H, Koch S, Granval P, Lecleire S, Charachon A, Barange K, Cesbron EM, De Widerspach A, Le Baleur Y, Barthet M, Poincloux L. Complete endoscopic sphincterotomy with vs. without large-balloon dilation for the removal of large bile duct stones: randomized multicenter study. Endoscopy. 2017 Oct;49(10):968-976. doi: 10.1055/s-0043-114411. Epub 2017 Jul 28. PMID 28753698